CLINICAL TRIAL: NCT06810791
Title: The Efficacy and Safety of Homoharringtonine Combined With Venetoclax and Azacitidine Versus Standard Chemotherapy or VA in the Treatment of Acute Myeloid Leukemia With High-risk, a Multicenter, Prospective, Randomized Study
Brief Title: HVA vs IA/DA or VA in the Treatment of ND HR-AML
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Guangdong Second Provincial General Hospital (Other); Jiangmen Central Hospital (Other); Shenzhen Second People's Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Dongguan People's Hospital (Other Government); First People's Hospital of Foshan (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Huizhou Municipal Central Hospital (Other); Shenzhen Hospital of Southern Medical University (Other); Affiliated Hospital of Guangdong Medical University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); First People's Hospital of Chenzhou (Other); Hunan Provincial People's Hospital (Other); Ganzhou City People's Hospital (Other); First Affiliated Hospital of Gannan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2024-576
Record Dates: First submitted 2025-01-16; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Newly Diagnosed Acute Myeloid Leukemia With High Risk
Keywords: HVA regimen; Intensive chenmotherapy; Fit; randomized controlled trial; Phase 3; VEN combined with AZA; Unfit; Newly diagnosed; High risk; Acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Patients with newly diagnosed AML with high risk will be divided into two cohorts, including patients being eligible for intensive chemotherapy and those with unfit status according to Ferrara 2013 criteria. In the fit cohort, patients will be randomized into accepting HVA versus IA/DA for induction with a ratio of 1:1. In the unfit cohort, patients will be randomized into accepting HVA versus VA for induction with a ratio of 1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IC regiment for Fit-AML (Active Comparator)
  Interventions: Drug: Standard Chemotherapy
- HVA regiment for Fit-AML (Experimental)
  Interventions: Drug: HVA
- VA regiment for unfit-AML (Active Comparator)
  Interventions: Drug: VA
- HVA regiment for unfit-AML (Experimental)
  Interventions: Drug: HVA

INTERVENTIONS:
Drug: HVA — Homoharringtonine (HHT) is given by venous drip daily at 1 mg/m2 from day 1 to 7. Venetoclax (VEN) is given 100 mg on day 1, 200 mg on day 2, and 400 mg orally from day 3 to day 14. Azacitidine (AZA) is given 75 mg/m2 subcutaneously from day 1 to 7.
  Arms: HVA regiment for Fit-AML; HVA regiment for unfit-AML
Drug: VA — VEN is given 100 mg on day 1, 200 mg on day 2, and 400 mg orally from day 3 to day 28, and AZA (75 mg/m2) is given subcutaneously from day 1 to 7.
  Arms: VA regiment for unfit-AML
Drug: Standard Chemotherapy — Standard Chemotherapy includes IA(Idarubicin combined with Cytarabine) or DA(Daunorubicin combined with Cytarabine). IDA is given by venous drip daily at 12mg/m2, or DNR is given by venous drip daily at 60mg/m2, from day 1-3, combined with Ara-C at 100mg/m2 by continuously venous drip from day 1-7.
  Arms: IC regiment for Fit-AML

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of homohartonine combined with venetoclax and azacitidine (HVA) versus intensive chemotherapy (IA/DA) or venetoclax combined with azacitidine (VA) in newly diagnosed high-risk AML patients.

DETAILED DESCRIPTION:
The HVA regimen exerts a synergistic pro-apoptotic effect and has demonstrated significant clinical efficacy against R/R AML and also overcomes adaptive resistance observed in the VA regimen. Exploratory work with small sample sizes in first-line settings suggests that combination of HHT and Ven+AZA exhibits potent anti-AML effects with good safety profiles, particularly in overcoming the impact of high-risk factors associated with AML relative to standard treatments. This indicates its potential as a more ideal option for the treatment of newly diagnosed AML with high risk factors. Therefore a prospective, multi-center, randomized controlled clinical study is planned to evaluate the efficacy and safety of the HVA regimen compared to intensive chemotherapy (IA/DA) or Venetoclax plus azacitidine (VA) regimens in newly diagnosed high-risk fit-AML or unfit AML patients.

ELIGIBILITY:
Inclusion Criteria:

* According to the world health organization (WHO) classification of newly diagnosed with AML patients;
* Age ≥18 years old;
* High-risk patients should meet any of the following criteria: ① High risk group according to the European Leukemia Risk stratification (ELN) 2022; (2) Secondary AML (sAML) which develops from myelodysplastic syndrome (MDS), bone marrow hyperplastic tumor (MPN) or chronic myeloid cell leukemia, et.; (3) Treatment-related AML (t-AML), Patients have a history of cytotoxic treatment record or ionizing radiation therapy.
* Patients did not receive anti-AML therapy (except leukopenia therapy, such as hydroxyurea or cytarabine < 1.0g/d) after the diagnosis of AML;
* Expected survival ≥12 weeks;
* The eastern tumor cooperation group (ECOG) score 3 points or less;
* Kidney function: creatinine clearance acuity 30 ml/min;
* Liver function: ALT < 5 times normal value, bilirubin < 3 times normal value;
* Sign the informed consent form and understand and abide by the plan calls for process.

Exclusion Criteria:

* Acute promyelocytic leukemia;
* With central nervous system leukemia (CNSL) ;
* The cardiac function > level 2;
* The AIDS virus (HIV) infection;
* Other clinical significance of uncontrolled condition, including but not limited to: (1) out of control, or active systemic infection (viruses, bacteria or fungi); (2) chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) requiring treatment; (3) need to actively deal with the merger of the second tumor;
* Can't take oral treatment or having a gastrointestinal disease impact ing the absorption;
* Being allergy to the experimental drugs;
* Pregnant and lactating women;
* Patients who could not understand or adhere to the study protocol;
* Patients deemed by the investigator to be ineligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 876 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CRc) | At the end of cycle 2 (each cycle is 28 days).
  CRc includes complete remission (CR) and complete remission accompanied with with incomplete count recovery (CRi).

SECONDARY OUTCOMES:
Complete remission (CR) | At the end of cycle 2 (each cycle is 28 days).
  Complete remission is defined as BM with >5% blasts and without extramedullary infltration and recovery of peripheral blood cells.
Overall response rate (ORR) | At the end of cycle 2 (each cycle is 28 days).
  ORR includes CRc, partial response (PR), and morphologic leukemia-free state (MLFS).
DOR | 1 year
  duration of response
Rate of Measurable residual disease (MRD) negative | At the end of cycle 2 (each cycle is 28 days).
  MRD is monitored using flow cytometric analysis with a positive MRD threshold of 0.1%.
Overall survival (OS) | 1 year
  OS is calculated from enrollment to death or the last follow-up.
Event-free survival (EFS) | 1 year
  EFS is calculated from enrollment to the date of relapse or death or the last follow-up.
Adverse events (AE) | The first dose until 28 days after treatment discontinuation
  AE are recorded from the first dose until 28 days after treatment discontinuation and are graded according to the NCI Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Guopan Yu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No